CLINICAL TRIAL: NCT05317221
Title: Developing Breast (Cancer) Organoids
Status: Recruiting | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other); Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: Organoids Breast
Record Dates: First submitted 2022-03-16; First posted 2022-04-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extra tube of blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: The is only 1 arm: all breast cancer patients undergoing surgery.
  Interventions: Other: Not an extra intervention, tissue taken in routine practice will be used.

INTERVENTIONS:
Other: Not an extra intervention, tissue taken in routine practice will be used. — No extra intervention: using tumour tissue taken during surgery in standard of care.

SUMMARY:
Currently, only a few validated biomarkers and models exist guiding or predicting treatment response for specific patient groups. Therefore, a patient-tailored clinical model needs to be developed to address tumour heterogeneity and thereby guide treatment selection on an individualized level. Organoids are patient-derived aggregates that grow in 3D and maintain self- renewal pluripotency and lineage-specific differentiation. Therefore, in contrast with conventional cell lines, they are thought to sustain patient heterogeneity and characteristics and are consequently already in use for drug response screening.

This now offers the opportunity to investigate if the primary patient breast cancer organoid platform reflects disease progression, treatment response and relapse in patients with different clinical breast cancer subtypes.

Goal: To develop a living biobank from prospective patient-derived breast cancer tissue. The questions we will address are:

1. Do patient-derived breast cancer organoids retain the clinical behaviour and characteristics of the primary patient tumour?
2. Can BC organoids be used to derive prognostic and predictive biomarkers to inform treatment decisions?
3. Can the investigators utilize BC organoids to discover novel actionable targets and combination treatments for therapeutic intervention for breast cancer patients?
4. Can BC organoids be used to discover mechanisms of treatment resistance and relapse?

DETAILED DESCRIPTION:
The investigators will select patients with a diagnosis of breast cancer who undergo breast surgery. Patients will be asked informed consent for the use of a small (0,2-1 cm3) sample of the excised breast tumour and the collection of a blood sample (6ml)for whole-exome sequencing (WES) to compare the genetic profile of the patients with the organoids and the patient biopsy. The patients will not undergo any additional treatment or procedure in addition to the planned routine procedure for the surgical resection of their primary breast tumour.

Patient will undergo standard diagnostic procedures and treatment according to the Dutch breast cancer surgery guidelines. After surgery, the pathologist will provide -after pathological diagnosis- rest (tumour) tissue from the resection to the lab. This material will then be used to develop breast cancer organoids. As part of the routine surgical procedure, 6 ml of blood will be collected. Participation in this study does not lead to additional actions other than reading the patient information and signing the informed consent. Therefore, participation does not change the patient's treatment or outcome.

ELIGIBILITY:
Inclusion Criteria:

* Female,
* >18 years,
* Family Anamneses
* Breast cancer (proven by histopathology), Included subtypes; (ER-,PR- HER2-); (ER+, PR+, HER2-); (ER+, PR+ HER2+).
* Primary surgery (lumpectomy or mastectomy)

Exclusion Criteria:

- Physically or mentally incapable or incompetent to sign informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All breast cancer patients that meet the criteria mentioned above.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Living biobank | 12 months
  The development of a patient derived breast cancer living biobank using 3D organoid technology reflecting the most prominent clinical subtypes.

SECONDARY OUTCOMES:
Organoids. | 12 months
  Cultivate breast cancer organoids that can be used to predict the treatment response to existing and novel combination treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Vooijs, PhD, Principal Investigator — Maastricht University; Marjolein Smidt, MD, PhD, Principal Investigator — Maastricht University Medical Center; Loes Kooreman, MD, Principal Investigator — Maastricht University Hospital (MUMC+); Maaike De Boer, MD, PhD, Principal Investigator — Maastricht University Hospital (MUMC+)
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands